CLINICAL TRIAL: NCT05814913
Title: Culturally Adapted Psychosocial Interventions for Early Psychosis in a Low-resource Setting: a Large Multi-center Randomised Controlled Trial
Brief Title: Culturally Adapted Psychosocial Interventions for Early Psychosis in a Low-resource Setting
Acronym: CaPSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL/CAMH-CaCBT+CulFI-002
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Psychosis
Keywords: First Episode Psychosis; LAMIC; Family Intervention; CBT; Paksitan
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers doing outcome assessment will be blind to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CaCBT for psychosis (Experimental): CaCBT is a culturally adapted psychosocial intervention for people with early psychosis that comprises of 12 sessions. These sessions are conducted individually on a weekly basis and last 45-60 minutes
  Interventions: Behavioral: CaCBT for psychosis
- CulFI Intervention (Experimental): CulFI is a culturally adapted psychosocial intervention delivered over 10 sessions of 40-60 minutes, weekly for the first 8 weeks and fortnightly for the remaining 4 weeks. Sessions are delivered to patients and their carers, though patient participation in sessions is not necessary.
  Interventions: Behavioral: Culturally adapted Family Intervention (CulFI) for psychosis
- Treatment as Usual (TAU) (No Intervention): TAU will be ascertained by the participant's treating physician. Research staff will record the nature and intensity of TAU delivered to each participant over a period of 3 months.

INTERVENTIONS:
Behavioral: CaCBT for psychosis — The CaCBT intervention is based on the intervention manual developed by David Kingdon and Douglas Turkington, and culturally adapted by our group. CaCBT aims to take a collaborative approach to gaining an understanding of the symptoms
  Arms: CaCBT for psychosis
Behavioral: Culturally adapted Family Intervention (CulFI) for psychosis — CulFI intervention comprises of Family psychoeducation; cognitive-behavioural skills training for stress-management, coping and problem solving; crisis intervention and suicide risk management; relapse prevention; education and support regarding the family environment, including communication training. The components are designed to facilitate an understanding about psychosis, the emotional impact of the illness on family relationships, to promote more adaptive coping strategies and minimize relapse risk.
  Arms: CulFI Intervention

SUMMARY:
Primary Aims:

To determine the clinical efficacy of Culturally adapted Cognitive Behavioral Therapy (CaCBT) and Culturally adapted Family Intervention (CulFI) compared to Treatment As Usual (TAU) on reducing overall symptoms of psychosis in patients with First Episode Psychosis (FEP) in Pakistan.

Secondary Aims:

1. To determine the efficacy of CaCBT and CulFI compared to TAU on positive and negative symptoms of psychosis, general psychopathology, depressive symptoms, quality of life, general functioning, and insight in patients with FEP in Pakistan.
2. To determine the efficacy of CaCBT and CulFI compared to TAU on improving carer experience, carer wellbeing, carer illness attitudes and symptoms of depression and anxiety in family and carers of patients with FEP in Pakistan.
3. To determine the comparative effect of CaCBT and CulFI in improving patient and carer related outcomes in individuals with FEP in Pakistan.
4. To estimate the economic impact of delivering culturally appropriate psychosocial interventions in low-resource settings
5. To explore delivery and reach of each intervention, tolerability of intervention components, acceptability of interventions, understanding mechanism of change and developing an understanding of barriers and facilitators to future adoption using process evaluation.

Study design and setting:

This will be a multi-centre, assessor masked, individual, three-arm randomised controlled trial (RCT).

Sample Size:

The study aims to recruit a total of N=390 participants with FEP

DETAILED DESCRIPTION:
Family Intervention (FI) and cognitive behavior therapy (CBT) are among the most efficacious psychosocial interventions to prevent relapse in schizophrenia. However, there is limited evidence from LMICs that supports the clinical efficacy and cost-effectiveness of delivering these psychosocial interventions to individuals with FEP. We aim to determine the clinical efficacy and cost-effectiveness of Culturally adapted Cognitive Behavioral Therapy (CaCBT) and Culturally adapted Family Intervention (CulFI) compared to TAU in reducing overall symptoms of psychosis in individuals with FEP in Pakistan. The study will include 390 participants with FEP from psychiatric units of hospitals and community settings in ten centres (i.e. Karachi, Lahore, Rawalpindi, Hyderabad, Qambar Shahdakot, Shaheed Benazirabad, Sukkur, Peshawar, Quetta and Multan).

Consented participants meeting eligibility criteria will be randomised in a 1:1:1 allocation to CaCBT + TAU, CulFI + TAU or TAU alone. Participants in CaCBT intervention group will receive 12-weekly one-to-one sessions. Participants in CulFI group will receive 10-weekly one-to-one sessions. Each CaCBT and CulFI session will last for approximately 1 hour. Sessions will be delivered by trained psychologists who will receive regular weekly supervision to maintain fidelity. Assessments will be carried out at baseline, months 3, 6, and 12 by trained, blinded assessors. . Process evaluation will help to build the implementation knowledge base for proposed interventions across study settings. We will conduct economic evaluations (i.e., the cost-effectiveness and cost-utility analyses) of the CaCBT and CulFI interventions, as add-on to TAU.

ELIGIBILITY:
Inclusion Criteria for patient participants:

* Individuals of all genders aged over 18 years; diagnosis of schizophrenia confirmed by Structured Clinical Interview for DSM (SCID) meeting DSM-5 criteria for schizophrenia, schizophreniform or schizoaffective psychosis
* Scored at least 4 on the PANSS delusions or hallucinations items, or at least 5 on suspiciousness, persecution, or grandiosity items
* stable on medication for the past four weeks
* in contact with mental health services
* within 3 years of diagnosis
* able to demonstrate the capacity to provide informed consent to take part in the study
* potential participants must have a carer or relative who is also willing to participate in the study to be eligible

Exclusion Criteria for patient participants:

* Active DSM-5 substance use disorder (except nicotine or caffeine) or dependence within the last three months
* A score of 5 or more on the PANSS conceptual disorganisation item
* Individuals who have received structured psychological intervention within the past 3 months
* Relevant CNS or other medical disorders that would impact participation
* Diagnosis of intellectual disability
* Unstable residential arrangements

Family member/Carer participant inclusion criteria:

* Living with or spending at least 10 hours per week in face-to-face contact with an individual with early psychosis and assuming a caring role
* Age>18 years
* Able to give informed written consent.

Family member/Carer participant exclusion criteria:

* Active DSM-5 substance use disorder
* Received psychological intervention within the past 3 months
* Unstable residential arrangements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | Change in scores from baseline to months 3, 6, and 12
  The PANSS is a structured interview use to evaluate the prevalence and severity of the positive, negative and general psychiatric symptoms of schizophrenia. The higher the score the greater symptoms severity. potential ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale.

SECONDARY OUTCOMES:
Calgary Depression Scale for Schizophrenia | Change in scores from baseline to months 3, 6, and 12
  The CDSS is a 9-items scale which evaluates depression in individuals with psychosis. The minimum score is 0 and maximum 30.Higher scores indicate greater depressive severity
EuroQol-5 Dimensions | Change in scores from baseline to months 3, 6, and 12
  EuroQol-5D (EQ- 5D) will be used to assess health-related quality of life over 5 dimensions (mobility, self-care, daily activities, pain-discomfort, anxiety and depression). Higher score indicates better quality of life.
World Health Organization Disability Assessment Scale | Change in scores from baseline to months 3, 6, and 12
  It is a self-administered questionnaire based on 36 items that measures health and disability. The scoring has three steps: Step 1 - Summing of recoded item scores within each domain. Step 2 - Summing of all six domain scores. Step 3 - Converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability
Schedule for Assessment of Insight | Change in scores from baseline to months 3, 6, and 12
  The Schedule for Assessment of Insight is used to evaluate the three different aspects of insight: treatment compliance, recognition of illness and re-labelling of psychotic phenomena
Experience of Caregiving Inventory | Change in scores from baseline to months 3, 6, and 12
  The ECI is a thorough measure that assesses the experiences of caring for a family member with severe mental illness
Carer Well-Being and Support | Change in scores from baseline to months 3, 6, and 12
  The CWS is an instrument to assess the wellbeing and support of a carer
Illness Perception Questionnaire | Change in scores from baseline to months 3, 6, and 12
  The IPQ is used to evaluate carer beliefs about schizophrenia
Generalized Anxiety Disorder | Change in scores from baseline to months 3, 6, and 12
  A 7-item scale measuring anxiety. Higher score indicates higher anxiety. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Patient Health Questionnaire (PHQ-9) | Change in scores from baseline to months 3, 6, and 12
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. PHQ-9 total score for the nine items ranges from 0 to 27. Higher score indicates greater depression severity
Cognitive Behaviour Therapy Rating Scale | Fidelity will be measured after completion of the intervention ( at 3rd month)
  Fidelity to the manuals of the interventions will be assessed via recorded sessions using Cognitive Behaviour Therapy Rating Scale
Cognitive Therapy for Psychosis Adherence Scale | Therapists' adherence will be measured after completion of the intervention ( at 3rd month)
  Therapists' adherence to the manuals of the interventions will be assessed via recorded sessions using Cognitive Therapy for Psychosis Adherence Scale
The Psychosocial Treatment Compliance Scale (PTCS) | Participants' compliance with psychosocial treatment will be assessed at end of intervention (3-months)
  This is a is a reliable and valid scale which is used to measure the compliance to psychosocial treatment of people with psychotic disorders
Treatment Adherence Rating Scale | Participants' adherence will be assessed at end of intervention at 3, 6 and 12 months
  This scale will be used to assess the antipsychotic medication adherence of participants
Session Attendance Log | Session attendance for each session for 3 months
  A session log will be maintained for each participant to maintain record of attendance for each session of assigned intervention.
The block design | Change in scores from baseline to 3, 6 and 12-month follow up
  The block design sub-test from the Wechsler Intelligence Scales will be sued to assess cognitive functioning. The higher score on the scale reflects better cognitive functioning
Matrix ReasoningTest | Change in scores from baseline to 3, 6 and 12 month follow up.
  The matrix reasoning sub-test from the Wechsler Intelligence Scales will be used to assess visual information processing and abstract reasoning skills. Higher scores on the scale indicate better visual information processing and abstract reasoning skills.
Picture Completion Test | Change in scores from baseline to 3, 6 and 12-month follow up
  The picture completion sub-test from the Wechsler Intelligence Scales measures measures visual perception, specifically, alertness to visual details. Higher score on this sub-scale indicate better cognitive skills in terms of visual perception.
Visual Puzzles Test | Change in scores from baseline to 3, 6 and 12-month follow up
  The Visual Puzzles sub-test from the Wechsler Intelligence Scales measures visual intelligence. Higher score on this sub-test indicates high visual intelligence.
The Oral Fluency test | Change in scores from baseline to 3, 6 and 12-month follow up
  This test measures the ability to evoke valid and distinct exemplars of a particular category. Higher score on this scale indicate better cognitive ability.
Memory for Design | Change in scores from baseline to 3, 6 and 12-month follow up
  The test examines visual recall of an individual. Higher score indicate better cognitive skills.
Coughlan Learning Task (verbal) | Change in scores from baseline to 3, 6 and 12-month follow up
  This test assesses verbal memory. Higher score on this test indicates better verbal memory.
Coughlan Learning Task (visual) | Change in scores from baseline to 3, 6 and 12-month follow up
  This test assesses visual memory. Higher score on this test indicates better visual memory.

CONTACTS AND LOCATIONS:
Overall Officials: Omair Husain, MD, Principal Investigator — Centre for Addiction and Mental Health; Imran B Chaudhry, MD, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Civil hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Husain MO, Khoso AB, Kiran T, Chaudhry N, Husain MI, Asif M, Ansari M, Rajput AH, Dawood S, Naqvi HA, Nizami AT, Tareen Z, Rumi J, Sherzad S, Khan HA, Bhatia MR, Siddiqui KMS, Zadeh Z, Mehmood N, Talib U, de Oliveira C, Naeem F, Wang W, Voineskos A, Husain N, Foussias G, Chaudhry IB. Culturally adapted psychosocial interventions (CaPSI) for early psychosis in a low-resource setting: study protocol for a large multi-center RCT. BMC Psychiatry. 2023 Jun 16;23(1):444. doi: 10.1186/s12888-023-04904-8. PMID 37328751